CLINICAL TRIAL: NCT04533516
Title: Effectiveness of 12-Weeks Inspiratory Muscle Training With Manual Therapy in Patients With COPD: Randomized Controlled Study
Brief Title: Additional Manual Therapy Over Inspiratory Muscle Training in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Manual therapy in COPD
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe; Muscle Weakness
Keywords: copd; manual therapy; inspiratory muscle therapy
MeSH Terms: conditions — Muscle Weakness; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy additional over Inspiratory muscle training (Experimental): Participants receive manual therapy protocol session three times a week for 12 weeks. The manual therapy protocol session lasts 30 minutes and included of the following manual therapy techniques: suboccipital decompression, gliding of the cervical vertebral articulations in the anterior/posterior direction, myofascial release of sternocleidomastoid and trapezius muscles, gliding of sternoclavicular joint in the anterior/posterior direction, myofascial release of intercostal muscles and paravertebral muscles, diaphragmatic release, rib raising, mobilization of scapulothoracic joint, and gliding of the thoracic vertebral articulations in the anterior/posterior direction. And all participants receive inspiratory muscle training.
  Interventions: Other: Manual therapy technics; Other: Inspiratory Muscle Training
- Inspiratory Muscle Training (Active Comparator): Participants receive only inspiratory muscle training by using Threshold Inspiratory Muscle Training device. Training load is 40% of the measured maximum inspiratory pressure, weekly. Participants receive inspiratory muscle training session for 30 min-per day, 7 days per week, for 12 weeks.
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Manual therapy technics — Manual therapy technics
  Arms: Manual Therapy additional over Inspiratory muscle training
Other: Inspiratory Muscle Training — Inspiratory Muscle Training

SUMMARY:
The benefits of inspiratory muscle training(IMT) in patients with chronic obstructive pulmonary disease(COPD) were reported.But in severe COPD patients, benefit from IMT may be limited.There is need for further research in new and complementary modalities to improve IMT efficiency in severe COPD patients.Manual therapy(MT) additional over IMT may be such a new approach that has not yet been investigated in COPD.

Aims: To investigate effects of MT additional over IMT on functional capacity,respiratory muscle strength,pulmonary function,dyspnea, fatigue and quality of life in severe COPD patients.

Methods: It was a prospective single-blind randomized trial. 40 patients with COPD in Global Initiative for Chronic Obstructive Lung Disease(GOLD) stage III-IV were included. Patients were randomly assigned to receive either MT additional over IMT at 40% of maximal inspiratory pressure(MIP)(n= 20) or only IMT(n= 20) for 12 weeks. MT group received MT during 12 weeks for 40 minutes additional to IMT. Pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, functional capacity using six minute walk test, dyspnea using Modified Medical Research Council(MMRC) dyspnea scale, fatigue using fatigue severity scale and quality of life using St. George's Respiratory Questionnaire(SGRQ) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease
* Being clinically stable
* Having FEV1/FVC ratio of ≤ 50% of the predicted value after bronchodilator drugs.

Exclusion Criteria:

* Having an acute bronchitis,
* Having a pneumonia,
* Having an exacerbation of COPD,
* Having thoracic spinal scoliosis,
* Having substantial chest wall deformity, or acute rib or vertebral fracture.
* Unable to perform the pulmonary function test because of cognitive or physical impairments.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-29 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Test | 12 weeks
  Before the pulmonary function test, all subjects rested to avoid fatigue. The lung function test including forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and vital capacity (VC) was performed in a seated position using a portable spirometer according to the American Thoracic Society guidelines.
respiratory muscle strength | 12 weeks
  For respiratory muscle strength, maximal inspiratory pressure (MIP), and maximal expiratory pressure (MEP) were evaluated using an electronic pressure transducer. MIP was measured at residual volume, and MEP was measured from total lung capacity.
6 minute walk test | 12 weeks
  6 minute walk test (6MWT) was applied to measure exercise capacity. The patient's heart rate, breathing frequency, and oxygen saturation were monitored with the pulse oximeter, and the values were recorded before and after the test. The distance was expressed both as metres.
Dyspnea perception | 12 weeks
  Dyspnea perception was assessed using the modified Medical Research Council (MMRC) dyspnea scale, Levels of dyspnea are graded 0 (absence of dyspnea during strenuous exercise), to 4 (dyspnea during daily activities).
Fatigue perception | 12 weeks
  Fatigue perception was assessed with Turkish version of Fatigue Severity Scale. A high score indicates increased fatigue intensity and the maximum score of the scale is 63.
St.George Respiratory Questionnaire | 12 weeks
  Quality of life was measured using the Turkish version of St.George Respiratory Questionnaire (SGRQ). It is a specific quality of life questionnaire for respiratory diseases. SGRQ consists of three subscale and 50 items; symptoms (8 items), activities (16 items), effects of the disease (26 items). Each subscale is scored ranging from 0 to 100 points. High scores indicate that worsened the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- İstinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided